CLINICAL TRIAL: NCT02853383
Title: Registry of COPD Patients Who Undergo Outpatient Treatment or Are Under Surveillance at Outpatient Polyclinic Healthcare Institutions of the Russian Federation in Moscow
Brief Title: Registry of COPD Patients From Outpatient Polyclinic Healthcare Institutions of the Russian Federation in Moscow
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Interregional Public Organization, Russian Respiratory Society (Other)
Responsible Party: Sponsor
Other Study IDs: RRS-001
Record Dates: First submitted 2016-07-14; First posted 2016-08-02 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Chronic Obstructive Pulmonary Diseases, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

SUMMARY:
To describe the clinical profile of COPD patient who is under outpatient surveillance at polyclinic institutions of Moscow (including demographic data (age, gender, ethnicity, occupation), smoking status, disease duration, disease severity grade, distribution by disease phenotype, disease exacerbation rate in the setting of real-life clinical practice).

DETAILED DESCRIPTION:
The registry of COPD patients in fact represents non-interventional multicenter retrospective study including all COPD patients included into the registry retrospectively from patients medical records and newly diagnosed under outpatient surveillance at the selected polyclinic institutions of Moscow.

The registry will include all patients with registered diagnoses J40 - J44 according to ICD-10 with spirometry results confirming COPD diagnosis, who are at the study start under outpatient surveillance, and also newly registered patients diagnosed with COPD (ICD-10 J40 - J44, as confirmed by spirometry results) during the conduction of the registry program at the selected polyclinic institutions of Moscow (according to ICD: J40 - Bronchitis, not specified as acute or chronic, J41 - Simple and mucopurulent chronic bronchitis, J41.0 - Simple chronic bronchitis, J41.8 - Mixed simple and mucopurulent chronic bronchitis, J 42 - Unspecified chronic bronchitis, J 43 - Emphysema, J 44 - Other chronic obstructive pulmonary disease) based on regular (yearly) retrospective analysis of patient records with data entry into a consolidated database.

It is planned to enrol into the study approximately 2000 male and female patients over 40 years of age with diagnosed COPD (as confirmed by spirometry results).

The present observational multicenter descriptive study will be conducted in the setting of routine clinical practice of outpatient polyclinic institutions. There is no hypothesis to be tested in this study.

The study will be conducted in outpatient polyclinic institutions of the primary medical care system of Moscow. Pulmonologists of the primary medical care system will be engaged as investigators. These are the physicians, whom the patients with tentative COPD diagnosis are referred to in the Russian Federation and who within the scope of their responsibilities have access to source medical records and who evaluate the quality of diagnosis and extent of treatment prescribed to COPD patients.

The present study is observational therefore it does not require a treatment regimen or directions for patient management. The patients receive medical care in line with routine practice for treatment of this disease in the Russian Federation. Patient participation in the study should not in any way affect the principles and extent of treatment received by the patient according to routine clinical practice.

Physicians-investigators will enter into the study the information (data) concerning COPD patients, both those already registered at the selected medical treatment and preventive care institution, and newly registered patients as they seek attention at the outpatient polyclinic institutions.

The main purpose of the present study consists in collection of data concerning COPD patients who under surveillance at outpatient polyclinic institutions of Moscow using patient medical records and their medical history. This protocol does not specify any obligatory visits or examinations.

Patient data will be entered into the registry de-identified. The patients will be identified by their screening number and initials. Then the Physician-investigator will evaluate patient compliance with inclusion criteria. The study will enrol patients meeting all the inclusion criteria and not having any of the exclusion criteria.

Only the physician who enters patient data into the regional COPD registry possesses patient contact information, and henceforth only this physician will enter de-identified patient data according to study design. This physician does not influence the choice of examination extent, treatment strategy and medication.

ELIGIBILITY:
Inclusion Criteria:

* smokers or ex-smokers, with previously diagnosed COPD
* COPD diagnosis corresponding to ICD codes J40 - J44 (J40 - Bronchitis, not specified as acute or chronic, J41 - Simple and mucopurulent chronic bronchitis, J41.0 - Simple chronic bronchitis, J41.8 - Mixed simple and mucopurulent chronic bronchitis, J 42 - Unspecified chronic bronchitis, J 43 - Emphysema, J 44 - Other chronic obstructive pulmonary disease
* COPD diagnosis confirmed by spirometry results (spirometry is performed as normal with bronchodilator testing using salbutamol 400 µg, post-BD FEV1\ FVC < 0.7)

Exclusion Criteria:

* Tuberculosis
* Sarcoidosis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Randomly selected polyclinic institutions of Moscow will take part in the study and enrol into the registry 2000 patients for representativeness of sample for analysis of COPD prevalence in Moscow.
  The patient population includes male and female patients over 40 years of age, smokers or ex-smokers, under outpatient surveillance at polyclinic institutions of Moscow with diagnosis codes according to ICD J40 - J44 and diagnosed COPD, as confirmed by spirometry results
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
COPD prevalence among patients registered in the healthcare system of Moscow (under outpatient surveillance at polyclinic institutions of Moscow). | 1 day
  COPD prevalence among patients registered in the healthcare system of Moscow (under outpatient surveillance at polyclinic institutions of Moscow).
To describe the clinical profile of COPD patient in Moscow (including demographic data (age, gender, ethnicity, occupation), smoking status, disease duration, disease severity grade | 1 day
  To describe the clinical profile of COPD patient who is under outpatient surveillance at polyclinic institutions of Moscow (including demographic data (age, gender, ethnicity, occupation), smoking status, disease duration, disease severity grade, distribution by disease phenotype, disease exacerbation rate in the setting of real-life clinical practice).

SECONDARY OUTCOMES:
Percentage of patients with different disease phenotypes among outpatients | 1 day
  Characterize percentage (%) of COPD patients wth different disease phenotypes among outpatients
Percentage of prescriptions of medicinal products to COPD patients depending on disease severity grade in the setting of real-life clinical practice | 1 year
  Percentage of prescriptions of medicinal products to COPD patients depending on disease severity grade in the setting of real-life clinical practice
Distribution (%) of COPD patients who seek attention from primary medical care physicians by severity of airway obstruction | 1 year
  Distribution (%) of COPD patients who seek attention from primary medical care physicians by severity of airway obstruction
Mean number of exacerbations requiring medical attention (outpatient prescription of oral corticosteroids and/or antibiotics) in the last year in COPD patients | 1 year
  Mean number of exacerbations requiring medical attention (outpatient prescription of oral corticosteroids and/or antibiotics) in the last year in COPD patients
Mean number of hospitalizations in the last year in COPD patients | 1 year
  Mean number of hospitalizations in the last year in COPD patients
Disease burden based on the collected data concerning the duration of temporary disability | 1 year
  Disease burden based on the collected data concerning the duration of temporary disability in days
Disease burden based on the collected data concerning the outpatient visits due to COPD | 1 year
  Disease burden based on the collected data concerning the outpatient visits due to COPD in last year
To determine the percentage of patients with eosinophilic inflammation according to haematology results | 3 years
  To determine the percentage of patients with eosinophilic inflammation according to haematology results
To describe treatment regimens prescribed to COPD patients depending on disease severity grade in the setting of real-life clinical practice | 3 years
  To describe treatment regimens prescribed to COPD patients depending on disease severity grade in the setting of real-life clinical practice
To establish the percentage of medical prescriptions for treatment of COPD patients which comply with current Federal clinical guidelines for diagnosis and treatment of chronic obstructive pulmonary disease. | 1year
  To establish the percentage of medical prescriptions for treatment of COPD patients which comply with current Federal clinical guidelines for diagnosis and treatment of chronic obstructive pulmonary disease.
To evaluate the disease burden based on the collected data concerning the duration of temporary disability of patients under outpatient surveillance | 1 year
  To evaluate the disease burden based on the collected data concerning the duration of temporary disability of patients under outpatient surveillance
To evaluate the disease burden based on the collected data concerning the number of hospitalizations due to COPD exacerbations | 1 year
  To evaluate the disease burden based on the collected data concerning the number of hospitalizations due to COPD exacerbations in last year

CONTACTS AND LOCATIONS:
Overall Officials: Andrey S Belevskiy, M.D., Ph.D., Principal Investigator — Interregional Public Organization "Russian Respiratory Society'
Locations (1):
- Russian respiratory Society, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT02853383/Prot_SAP_000.pdf